CLINICAL TRIAL: NCT00700167
Title: Immune Responses To Antigen-Bearing Dendritic Cells in Patients With Malignancy - A Phase I Trial in Melanoma
Brief Title: Immune Responses To Antigen-Bearing Dendritic Cells in Patients With Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Rockefeller University (Other)
Responsible Party: James Young, M.D, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-098; NIH CA33049
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Melanoma
Keywords: ANTIGENBEARING DENDRITIC CELLS; 98-098
MeSH Terms: conditions — Melanoma

ARMS (1):
- 1 (Experimental): The vaccine will be split between as many as 10 injections, more or less. Each shot will be about 1/25th to 1/50th of a teaspoon (100 to 200 microliters). Each vaccine will be injected with a tiny needle just under your skin. This will usually cause a very small area of swelling at the injection site that may last for a few minutes to an hour or so. You will receive two additional "booster" doses of the same vaccine every 4-6 weeks. This would mean that you receive a total of three vaccines over about 2-3 months.
  The vaccines will be given during an outpatient visit. If for some reason, you happen to be in the hospital, you can still receive the vaccines. These visits should take no longer than 15-30 minutes.
  Interventions: Biological: dendritic cell vaccine

INTERVENTIONS:
Biological: dendritic cell vaccine — The vaccine will be split between as many as 10 injections, more or less. Each shot will be about 1/25th to 1/50th of a teaspoon (100 to 200 microliters). Each vaccine will be injected with a tiny needle just under your skin. This will usually cause a very small area of swelling at the injection site that may last for a few minutes to an hour or so. You will receive two additional "booster" doses of the same vaccine every 4-6 weeks. This would mean that you receive a total of three vaccines over about 2-3 months.

SUMMARY:
Cancer cells make proteins called antigens that act as markers for the tumor cells. These antigens cannot cause the cancer itself. Special white blood cells, called T cells or T lymphocytes, recognize and respond to antigens. In many diseases, these and other cells in the immune system help your body get rid of the disease. However, T cells are normally resting, and they need other proteins on the diseased cell surface to begin working. Unfortunately, cancer cells do not usually make all the other proteins that T cells need to work. Therefore, T cells do not normally work against the cancer cells. We think this is one of the reasons that cancers grow and are not rejected by the body in the first place.

Another white blood cell, called a dendritic cell, does have most if not all of the special proteins needed to make T cells work to destroy cancer cells. However, dendritic cells do not normally have the cancer proteins on their surface. The challenge then is to combine the cancer markers (antigens) with these dendritic cells to make a vaccine. We think that the body's T cells might then react against the tumor and help destroy it. This study will see if putting tumor antigens made in a lab onto dendritic cells will make T cells work against tumor cells. We want to answer this question by injecting you with dendritic cells loaded with the antigens. Then we will check for a response based on lab studies and your own clinical course. We will compare your response against melanoma with your response against a common antigen, to which almost everyone has already been exposed. Flu, for example, is a common antigen to which most people have been exposed. We also need to test your response to an antigen that your body has not likely seen before. For example, we plan to use KLH (keyhole limpet hemocyanin), which is a pigment or color protein made from a sea creature known as a keyhole limpet. Each of these, the flu and KLH antigens, which should be harmless to you, will be used along with the dendritic cell-tumor vaccine. This will help us find out if the vaccine is working, based on the lab studies we will check before and after the vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic melanoma, AJCC stage III or IV, with histologic confirmation by Dept. of Pathology at MSKCC.
* Patients must be HLA-A*0201 positive.
* Expected survival of greater than 3 months.
* Karnofsky performance status 70 or better.
* Patients may not have received chemotherapy, immunotherapy, or radiation within approximately 4 weeks (approximately 6 weeks for nitrosoureas or mitomycin) before participation in this protocol.
* Patients should not be receiving immune modifying pharmacologics (e.g., interferon) for approximately 2-4 weeks before enrollment.

Exclusion Criteria:

* Pregnant (clinically documented or positive pregnancy test within approximately 2 wks of study entry) or lactating women, because immunization will include differentiation antigens shared by melanoma tumors and melanocytes, and immune responses to these differentiation antigens could have unknown developmental sequelae to a fetus or infant.

Pregnancy tests are not required for post-menopausal women, and post-menopausal status by patient report should be documented accordingly.

* Patients requiring systemic corticosteroids or comparable exogenous immunosuppressive agent(s) (no exclusion for use of NSAIDs)
* Patients who have a known immunodeficiency (e.g., infection with HTLV-1,2, HIV-1,2; etc.) because of the T cell defects that would alter their responses and the investigators' ability to assess their outcomes accurately.
* Patients with preexisting retinal or choroidal eye disease.
* Patients with coexisting autoimmune diseases, except vitiligo.
* Patients with significantly impaired hematologic, hepatic, or renal function, e.g., ANC <1000, hgb < 8.0 g/dl, plts < 50,000/ul, AST >3x ULN, creatinine >2.0 or Cl creat <30ml/min, all assessed within approximately two weeks of study entry.
* Patients with serious coexisting medical illness.
* Patients with organ allografts.
* Patients who are s/p splenectomy or s/p splenic irradiation.
* Patients with active brain metastases.
* Patients with organic brain syndrome or psychologic impairment that would preclude participation and compliance with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2001-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and toxicity of immunizations of patients with stage III/IV melanoma, using autologous DCs pulsed with antigenic peptides expressed by melanoma, together with class I MHC (influenza) and class II MHC (KLH) -restricted control antigens. | conclusion of the study
Evaluate further the immunogenicity of tumor antigen-bearing dendritic cells, based on the same in vitro assays as above, measured pre-& post-dendritic cell immunization with the optimal biologic dose of DCs selected in the phase Ia portion of the trial. | conclusion of the study

SECONDARY OUTCOMES:
Is to monitor local DTH responses in vivo against the antigen-loaded DCs after booster immunizations. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: James Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Romano E, Rossi M, Ratzinger G, de Cos MA, Chung DJ, Panageas KS, Wolchok JD, Houghton AN, Chapman PB, Heller G, Yuan J, Young JW. Peptide-loaded Langerhans cells, despite increased IL15 secretion and T-cell activation in vitro, elicit antitumor T-cell responses comparable to peptide-loaded monocyte-derived dendritic cells in vivo. Clin Cancer Res. 2011 Apr 1;17(7):1984-97. doi: 10.1158/1078-0432.CCR-10-3421. Epub 2011 Feb 25. PMID 21355077
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org